CLINICAL TRIAL: NCT05151835
Title: A Novel Robotic Surgical System for Minimally Invasive Surgery: A Prospective, Single Center, Multi-speciality Study
Brief Title: Novel Robotic Surgical System for Minimally Invasive Surgery
Acronym: K2robo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan CHIU, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2021.472
Record Dates: First submitted 2021-11-05; First posted 2021-12-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Robotic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic Surgery (Experimental): Prospective single arm study to investigate effect of a novel robotic surgical system on safety, efficacy and outcomes for performance of minimally invasive surgery across urology, upper and lower GI surgery.
  Interventions: Device: K2 Robotic Surgical System

INTERVENTIONS:
Device: K2 Robotic Surgical System — The K2 Robotic Surgical System is a software-controlled, electro-mechanical system designed for surgeons to perform minimally invasive surgery in the thorax and abdomen. The K2 Robotic Surgical System consists of a Surgeon Console [SGC], a Patient Side Robot [PSR], and a Vision Cart [VCT], and is used with an endoscope, Surgical Instruments [SGI], and Accessories [ACC]. The surgeon views the three-dimensional endoscopic image on a High-Resolution Stereo Viewer (3D Viewer), which provides a view of the abdominal cavity and surgical instrumentation, along with icons and other user interface features.

SUMMARY:
This is a prospective single center cohort study on effect of a novel robotic surgical system for performance of minimally invasive surgery in multiple specialties. The targeted procedures include Urological, upper and lower GI robotic surgeries and the expected sample size will be 20 patients. The clinical outcomes for assessment include background demographics, operative time, perioperative complications as well as completion rate of procedure, hospital stay and recovery.

DETAILED DESCRIPTION:
This is a prospective single center cohort study on effect of a novel robotic surgical system for performance of minimally invasive surgery in multiple specialties. The targeted procedures include Urological, upper and lower GI robotic surgeries and the expected sample size will be 20 patients. The procedures will be standardized according to previously reported. The diseases for robotic surgical treatment will include prostate carcinoma, colorectal carcinoma, as well as esophageal hiatal diseases and gastric carcinoma. The clinical outcomes for assessment include background demographics, operative time, perioperative complications as well as completion rate of procedure, hospital stay and recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index <35 kg/m2
2. Suitable for the listed minimally invasive surgical procedures for treatment of respective diseases
3. Willingness to participate as demonstrated by giving informed consent

Exclusion Criteria:

1. Contraindication to general anesthesia
2. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic intervention
3. Untreated active infection
4. Noncorrectable coagulopathy
5. Presence of another malignancy or distant metastasis
6. Emergency surgery
7. Vulnerable population (e.g. mentally disabled, pregnancy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion to ordinary laparoscopic surgery of robotic surgical procedures performed using the novel K2 Robotic Surgical System | 30 days
  Rate of conversion to ordinary laparoscopic surgery of robotic surgical procedures performed using the novel K2 Robotic Surgical System is defined as the need to change to laparoscopic surgery during the procedure.

SECONDARY OUTCOMES:
Rate of perioperative complications | 30 days
  intraoperative complications and all complications occurring during the hospital stay or within 30 days after discharge will be graded according to the Clavien-Dindo classification
intraoperative time | 30 days
  Intraoperative Time
Blood Loss | 30 days
  Amount of blood loss in mls
Pain scores on a visual analog scale | 30 days
  Pain score in visual analog scale scoring system (minimum 0 and maxium 10, higher score represents more pain)
Analgesic requirement | 30 days
  Total dose of analgesic (Pethidine) used
Length of Hospital Stay | 30 days
  Days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Outside of US & Canada, China

IPD SHARING:
Plan to Share IPD: No